CLINICAL TRIAL: NCT05299970
Title: Effect of Fermented Millet Porridge on Gut Microbiota Diversity and Inflammation Markers in Women of Reproductive Age in Rural Burkina Faso: A Pilot Study
Brief Title: Fermented Millet Porridge, Gut Microbiota and Inflammation Status in Women
Acronym: LAFIABAGA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institut de Recherche en Sciences de la Sante, Burkina Faso (Other Government)
Collaborators: University Ghent (Other); Bill and Melinda Gates Foundation (Other)
Responsible Party: Principal Investigator, Laeticia Celine Toe, Principal Investigator, Institut de Recherche en Sciences de la Sante, Burkina Faso
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: NUT_IRSS_0001
Record Dates: First submitted 2022-03-20; First posted 2022-03-29 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Inflammation; Microbiome, Human
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- fermented porridge (Experimental): this study arm participant will consume fermented millet porridge, daily
  Interventions: Other: Fermented porridge
- Non-fermented porridge (Active Comparator): this study arm participants will consume non-fermented millet porridge, daily
  Interventions: Other: Fermented porridge

INTERVENTIONS:
Other: Fermented porridge — A millet porridge (fermented or not, depending on group allocation) serving will be provided to participants daily, for consumption. consumption will be directly observed.

SUMMARY:
Maternal undernutrition concerns 10-19% of women of reproductive age globally, the vast majority of which live in sub Saharan Africa and south Asia. Recommendations for nutritional interventions to tackle the problem range from per-pregnancy supplementation to upstream interventions targeting women of reproductive age before conception. To render the latter interventions cost-effective and sustainable, experts recommend to focus on food processing that leads to an enhanced nutrient content. One such method, which has been known and practiced for centuries in diverse societies, is fermentation. Traditionally fermented foods are diverse, widespread and highly appreciated in Burkina Faso. The present study aims to investigate the effect of fermented millet porridge on gut microbiota diversity, stool short chain fatty acid concentration and inflammation markers level in women of reproductive age living in rural Burkina Faso.

ELIGIBILITY:
Inclusion Criteria:

Participant are

* 18 to 49 years old
* Resident in the study area and do not plan to move within 5 months following the start of the study
* Are not on antibiotic treatment on inclusion and have not been in the previous 3 weeks.
* Do not suffer from any pathology that could interfere with their diet.
* Have no known allergy to pearl millet or its derivatives
* Agree to sign a consent to participate in the study-

Exclusion Criteria:

* Women under 18 or over 49
* Women not consuming pearl millet porridge due to allergy or food preference
* Women planning to move from the study area within 5 months of the start of the study
* Women with serious illnesses that may interfere with their diet
* Women on antibiotic treatment or at the time of inclusion or having been in the previous 3 weeks.
* In addition, women who will benefit from antibiotic therapy during the study will be excluded from the analysis

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 80 (Estimated)
Dates: Start 2022-03-21 (Actual); Primary Completion 2024-01-30 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
Gut microbiota diversity | 0 to 13 weeks
  gut microbiota alpha and beta diversity
Concentration of inflammation markers in blood and stool | 0 to 13 weeks
  Concentration of IL1-beta, IL 8, IL 6, IL 33, TNF-alpha, lipocalin 2, myeloperoxidase, calprotectin

SECONDARY OUTCOMES:
Concentration of short chain fatty acid in stool | 0 to 13 weeks
  Concentration of C2-C8 fatty acids in stool
concentration of macronutrients in millet dough and porridge | 2 to 8 weeks
  Levels of carbohydrates, lipids, protein, dietary fiber and phytates
relative abundance of bacterial and fugal micro-organisms in millet dough and porridge | 2 to 8 weeks
  Count of microbial populations
Concentration of Ferritin in plasma | 0- to 13 weeks
  Ferritin levels in Plasma
Number of participant with anemia | 0 to 13 weeks
  hemoglobin concentration in grams per deciliter

CONTACTS AND LOCATIONS:
Overall Officials: Laeticia C TOE, Principal Investigator — IRSS-DRO
Locations (1):
- IRSS-DRO, Bobo-Dioulasso, Houet, Région Des hauts-Bassins, Burkina Faso

IPD SHARING:
Plan to Share IPD: Yes
Data sharing plans will be done according to the BMGF policy
Supporting Information: CSR, Analytic Code